CLINICAL TRIAL: NCT07278466
Title: The COMParing App Support Strategies Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-1444; Protocol Version 9/26/2025 (Other: UW Madison); EDUC/COUNSELING PSYCH (Other: UW Madison); 1R01MH139512-01 (NIH)
Record Dates: First submitted 2025-12-02; First posted 2025-12-12 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Depression, Anxiety
Keywords: HMP app; healthy minds program; Microsupport; meditation
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Introductory Coaching (Experimental)
  Interventions: Other: Introductory Coaching Session
- Introductory Coaching with On-Demand email support (Experimental)
  Interventions: Other: Introductory Coaching Session; Other: On-Demand Email Support
- Introductory Coaching and microsupport (Experimental)
  Interventions: Other: Introductory Coaching Session; Other: Microsupport
- Introductory Coaching with On-Demand email support and microsupport (Experimental)
  Interventions: Other: Introductory Coaching Session; Other: On-Demand Email Support; Other: Microsupport
- Introductory Information (Experimental)
  Interventions: Other: Introductory Information Session
- Introductory Information with On-Demand email support (Experimental)
  Interventions: Other: Introductory Information Session; Other: On-Demand Email Support
- Introductory Information and microsupport (Experimental)
  Interventions: Other: Introductory Information Session; Other: Microsupport
- Introductory Information with On-Demand email support and microsupport (Experimental)
  Interventions: Other: Introductory Information Session; Other: On-Demand Email Support; Other: Microsupport

INTERVENTIONS:
Other: Introductory Coaching Session — Participant is randomized to receive a 30-minute meditation coaching session
  Arms: Introductory Coaching; Introductory Coaching and microsupport; Introductory Coaching with On-Demand email support; Introductory Coaching with On-Demand email support and microsupport
Other: Introductory Information Session — Participant is randomized to receive a 30-minute information session
  Arms: Introductory Information; Introductory Information and microsupport; Introductory Information with On-Demand email support; Introductory Information with On-Demand email support and microsupport
Other: On-Demand Email Support — email support throughout the 4 week intervention period
  Other Names: email
  Arms: Introductory Coaching with On-Demand email support; Introductory Coaching with On-Demand email support and microsupport; Introductory Information with On-Demand email support; Introductory Information with On-Demand email support and microsupport
Other: Microsupport — Text message microsupport throughout the 4 week intervention period
  Other Names: text message
  Arms: Introductory Coaching and microsupport; Introductory Coaching with On-Demand email support and microsupport; Introductory Information and microsupport; Introductory Information with On-Demand email support and microsupport

SUMMARY:
The overall purpose of this study is to help determine how best to incorporate small amounts of human and digital support into a meditation app. The meditation app used is the Healthy Minds Program (HMP) which provides training in four pillars of well-being (Awareness, Connection, Insight, Purpose) through a combination of podcast-style didactic material and guided meditation practices.

DETAILED DESCRIPTION:
Participants will be randomly assigned to various support conditions that vary across three binary factors,

1. Introductory coaching session vs introductory information session
2. On-demand email support (Yes/No)
3. Microsupport messages (Yes/No)

Participants will be screened for eligibility using a web-based screener that assesses inclusion and exclusion criteria. Eligible participants will receive a study overview and will have the option to go through an online consent process. After giving consent, participant will receive a text message to assess their ability to receive text messages and tab on a link embedded in the text message. Those who failed to go through this process will be screened out.

Participants consented will complete a baseline survey consisting of a series of questionnaires and daily check-in assessment sent to their phone. Only those who successfully complete the baseline survey and the first daily check-in survey will advance in the study. Participants will schedule a meeting with our study staff member after completing the baseline survey and first daily check-in survey. They will be assessed through questionnaires at baseline, weekly during the 4-week intervention period, and at 6-month follow-up. They will also complete daily check-in survey twice a day throughout the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Elevated symptoms of depression and/or anxiety (PHQ-9 greater than or equal to 10, GAD-7 greater than or equal to 10)
* Proficiency in English
* Access to a smartphone and internet
* Ability to receive text messages

Exclusion Criteria:

* Non-US citizen or legal resident (green card holder)
* History of psychosis or mania
* Suicidal ideation or thoughts of self-harm indicated by PHQ9 item 9 and BDI item 9
* Individuals who do not provide the information required for GUID generation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 688 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2029-01-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire Anxiety and Depression Scale (PHQ-ADS) Score | baseline, week 1, week 2, week 3, week 4, 6-month follow up
  The PHQ-ADS is scored by summing responses to its 16 items (combining the PHQ-9 and GAD-7), with scores ranging from 0 to 48, where higher scores indicate greater distress. Each item uses a 0-3 scale (0=Not at all, 3=Nearly every day). Common interpretation is 10 (mild), 20 (moderate), and 30 (severe) distress.

SECONDARY OUTCOMES:
Perceived Stress Scale (PSS) Score | baseline, week 1, week 2, week 3, week 4, 6-month follow up
  The Perceived Stress Scale is a 10-item scale where participants report their level of perceived stress (e.g., "In the last month, how often have you felt nervous and 'stressed'?"). It is scored on a 5-point Likert scale where 0 is "never" and 4 is "very often." Total scores range from 0 to 40 where higher scores indicate greater perceived stress.
PROMIS Toolbox Meaning and Purpose Score | baseline, week 1, week 2, week 3, week 4, 6-month follow up
  The PROMIS / NIH Toolbox Meaning and Purpose is a computer-adaptive measure where participants report how much meaning and purpose they experience in life (e.g., "I understand my life's meaning"). It is scored on a 5-point Likert scale where 1 = strongly disagree to 5 = strongly agree. It provides total scores as T-scores (mean = 50, SD = 10) where higher scores indicate more meaning and purpose in life.
NIH Toolbox Loneliness Score | baseline, week 1, week 2, week 3, week 4, 6-month follow up
  The NIH Toolbox Loneliness is a 5-item questionnaire where participants report how often in the past week they have felt loneliness. It is scored on a 5-point Likert scale where 1 = never to 5 = always. The total possible range of scores is 5-25 where higher scores indicate a greater sense of loneliness.
Beck's Depression Inventory (BDI) Item 9 Score | baseline, week 1, week 2, week 3, week 4, 6-month follow up
  scored from 0 (no suicidal thoughts) to 3 (severe suicidal thoughts)
Five Facet Mindfulness Questionnaire (Awareness subscale) Score | baseline, week 1, week 2, week 3, week 4, 6-month follow up
  The Five Facet Mindfulness Questionnaire Acting with Awareness Subscale is a 8-item subscale where participants report on their general ability to focus. It is scored on a 5-point Likert scale where 1 = never or very rarely true to 5 = very often or always true. The total possible range of scores is 8-40 where higher scores indicate a greater ability to focus.
Experiences Questionnaire Decentering subscale Score | baseline, week 1, week 2, week 3, week 4, 6-month follow up
  The Decentering subscale of the Experience Questionnaire is an 11-item questionnaire where participants report on their ability to decenter from their experience. It is scored on a 5-point Likert scale where 1 = never to 5 = all the time. The total possible range of scores is 11-55 where higher scores indicate a greater ability to decenter from experience.
Perseverative Thinking Questionnaire (PTQ) Score | baseline, week 4, 6-month follow up
  The PTQ is a self-report instrument assessing repetitive and uncontrolled thinking by asking participants to rate 15 items about the frequency, duration, and perceived uncontrollability of repetitive thoughts on a scale of 0-4. Scores range from 0 to 60. The higher the score, the higher the level of perseverative thinking or repetitive thoughts experienced by the individual.
Healthy Minds Index (HM Index) - Awareness Score | baseline, week 4, 6-month follow up
  The HM Index is a 17-item questionnaire assessing qualities trained in the HMP app (awareness, connection, insight, purpose). It is scored on a 0- to 4-point Likert scale where 0 = a low amount (e.g., never, not at all, none of the time) and 4 = a higher amount (e.g., always, to the highest degree, all of the time) of a particular quality. Total scores for the Awareness subscale is 0 to 16 where higher scores indicate more awareness.
Healthy Minds Index (HM Index) - Connection Score | baseline, week 4, 6-month follow up
  The HM Index is a 17-item questionnaire assessing qualities trained in the HMP app (awareness, connection, insight, purpose). It is scored on a 0- to 4-point Likert scale where 0 = a low amount (e.g., never, not at all, none of the time) and 4 = a higher amount (e.g., always, to the highest degree, all of the time) of a particular quality. Total scores for the Connection subscale range from 0 to 24, where higher scores indicate more connection.
Healthy Minds Index (HM Index) - Insight Score | baseline, week 4, 6-month follow up
  The HM Index is a 17-item questionnaire assessing qualities trained in the HMP app (awareness, connection, insight, purpose). It is scored on a 0- to 4-point Likert scale where 0 = a low amount (e.g., never, not at all, none of the time) and 4 = a higher amount (e.g., always, to the highest degree, all of the time) of a particular quality. Total scores for the Insight subscale range from 0 to 12, where higher scores indicate more insight.
Healthy Minds Index (HM Index) - Purpose Score | baseline, week 4, 6-month follow up
  The HM Index is a 17-item questionnaire assessing qualities trained in the HMP app (awareness, connection, insight, purpose). It is scored on a 0- to 4-point Likert scale where 0 = a low amount (e.g., never, not at all, none of the time) and 4 = a higher amount (e.g., always, to the highest degree, all of the time) of a particular quality. Total scores for the Purpose subscale range from 0 to 16, where higher scores indicate more purpose.
Growth Mindset Scale Adapted for Well-being Score | baseline, week 4, 6-month follow up
  The Wellbeing Growth Mindset scale is a 3-item scale where participants report whether they believe wellbeing is malleable (e.g., "Your well-being is something about you that you can't change very much."). It is scored on a 6-point Likert scale where 1 is "strongly disagree" to 6 being "strongly agree." Total scores range from 3 to 18 where higher scores indicate greater wellbeing growth mindset.
Digital Working Alliance Inventory (DWAI) Score | week 1, week 2, week 3, week 4
  DWAI is a six-item questionnaire designed to assess the working alliance within the Healthy Minds Program (HMP) app. It measures the user's connection and agreement with the app, focusing on the bond, tasks, and goals of the therapeutic relationship. It is scored on a 7-point Likert scale, with scores ranging from 6-42. Higher scores indicate a stronger working alliance with the HMP app.
Morning Daily Diary Items | Daily through the Intervention Period (up to 4 weeks)
  Morning daily diary will include single-item measures of mindfulness, decentering, connection, purpose, depression, anxiety, happiness, energy, stress, busyness, rumination (2 items), sleep quality, motivation to practice meditation, and expectations and challenges related to using the HMP. Each item will be rated on a 5-point Likert scale (1 = not at all, 5 = very much). Higher scores indicate greater levels of the respective construct, such as higher mindfulness, greater decentering, stronger sense of purpose, greater happiness, more severe depression or anxiety, better sleep quality, or greater motivation and perceived helpfulness or frustration with HMP use that morning. Daily means with and standard deviations will be reported.
Evening Daily Diary Items | Daily through the Intervention Period (up to 4 weeks)
  Evening daily diary will include single-item measures of mindfulness, decentering, connection, purpose, depression, anxiety, happiness, energy, happy event, stress exposure, rumination (2 items), and expectations related to using the HMP. Each item will be rated on a 5-point Likert scale (1 = not at all, 5 = very much). Higher scores indicate greater levels of the respective construct, such as higher mindfulness, greater decentering, stronger sense of purpose, more severe depression or anxiety, happy event and stressor exposure experience, or greater motivation and perceived helpfulness with HMP use that day. Daily means with and standard deviations will be reported.
Percentage of participants with a formal practice | Daily through the Intervention Period (up to 4 weeks)
  Participants' engagement in formal mindfulness practice will be assessed twice a day with a binary yes/no response. Formal practice is defined as using the HMP app.
Percentage of participants with an informal practice | Daily through the Intervention Period (up to 4 weeks)
  Participants' engagement in informal mindfulness practice will be assessed twice a day with a 5-point Likert scale (1 = not at all, 5 = all day long). Informal practice is defined as applying well-being practices in daily life.
Percentage of participants who received a text message and applied a well-being strategy | Daily through the Intervention Period (up to 4 weeks)
  Participants will indicate whether they received a text message from the study that day (yes/no). If they respond "yes," they will then report whether the message encouraged them to apply a wellbeing strategy (yes/no) and rate the extent to which they applied the strategy in their day-to-day activities on a 5-point Likert scale (1 = not at all, 5 = very much).
Extent to which participants applied a well-being strategy in their day-to-day activities | Daily through the Intervention Period (up to 4 weeks)
  Participants who received a text message and applied a well-being strategy will be asked to rate the extent to which they applied the strategy in their day-to-day activities on a 5-point Likert scale (1 = not at all, 5 = very much).

CONTACTS AND LOCATIONS:
Overall Officials: Simon Goldberg, PhD, Principal Investigator — UW Madison
Locations (1):
- Center for Healthy Minds, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF

REFERENCES:
- See also: Center for Healthy Minds — https://centerhealthyminds.org/